CLINICAL TRIAL: NCT01337635
Title: Treatment Of Vitamin D Deficiency And Effect On Atopic Dermatitis Severity
Brief Title: Vitamin D Deficiency and Atopic Dermatitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not meeting enrollment goals.
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, Yvonne Chiu, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHW 10/146, GC 1169
Record Dates: First submitted 2010-11-03; First posted 2011-04-19 (Estimated); Results first posted 2015-04-08 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Atopic Dermatitis; Vitamin D Deficiency
MeSH Terms: conditions — Dermatitis, Atopic; Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard dose vitamin D (Active Comparator): Treatment with cholecalciferol 400 IU daily at home.
  Interventions: Drug: Vitamin D
- High dose vitamin D (Active Comparator): Treatment with ergocalciferol 300,000 IU (6 capsules of 50,000 IU) as a single oral dose observed in clinic.
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Ergocalciferol 300,000 IU single oral dose Cholecalciferol 400 IU orally every day for 6 weeks

SUMMARY:
Atopic dermatitis is a chronic skin disease characterized by a defective skin barrier, inflammation, and increased propensity for skin infections. Vitamin D is a fat-soluble vitamin that is primarily acquired through local production in the skin after ultraviolet light exposure but can also be obtained through natural and supplemental dietary sources. This randomized controlled trial will examine the effects of vitamin D repletion on atopic dermatitis severity in patients with diagnosed deficiency. The investigators hypothesize that pediatric patients with moderate or severe atopic dermatitis and vitamin D deficiency will have improved cutaneous disease after treatment with high dose as compared to standard dose vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* Serum 25-hydroxyvitamin D level <20 ng/ml (<50 nmol/L)
* Diagnosed with atopic dermatitis by a CHW pediatric dermatologist
* Age 1-18 years old
* Primary residence in Milwaukee County
* Moderate and severe atopic dermatitis (Severity Scoring of Atopic Dermatitis [SCORAD] score greater than 15)
* On clinic protocol treatment for their atopic dermatitis (desonide ointment twice daily for the face and groin, triamcinolone 0.1% ointment twice daily for other areas)

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Chiu, MD, Principal Investigator — Children's Hospital and Health System Foundation, Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Dose Vitamin D | High Dose Vitamin D
Started | 3 | 4
Completed | 3 | 3
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Standard Dose Vitamin D: Treatment with cholecalciferol 400 IU oral daily at home for 6 weeks
- Total: Total of all reporting groups
Arm/Group | Standard Dose Vitamin D | High Dose Vitamin D | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 4 | 7
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 9 [3 to 15] | 5 [2 to 10] | 6.7 [2 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Atopic Dermatitis Severity at the Completion of Treatment
Description: SCORAD at the 6 week study visit. The SCORAD (SCORing Atopic Dermatitis) is a clinical tool used to assess the extent and severity of eczema. The SCORAD is scored 0-103, with a higher score indicating more severe atopic dermatitis (worse outcome).
Time Frame: 6 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Standard Dose Vitamin D | High Dose Vitamin D
Number analyzed (Participants) | 3 | 3
score on a scale | 33.1 [25.6 to 43.4] | 15.5 [3.5 to 30.2]

2. Secondary Outcome: Time to Restart Topical Steroids
Description: The time to restart topical steroids.
Time Frame: 6 weeks
Measure: Mean (Full Range); unit: days
Arm/Group | Standard Dose Vitamin D | High Dose Vitamin D
Number analyzed (Participants) | 3 | 3
days | NA [NA to NA] — No subjects restarted topical steroids during the study period. | NA [NA to NA] — No subjects restarted topical steroids during the study period.

ADVERSE EVENTS:
Arm/Group | Standard Dose Vitamin D | High Dose Vitamin D
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No